CLINICAL TRIAL: NCT06888115
Title: Phase I Clinical Study to Evaluate the Pharmacokinetics and Safety of CS0159 Tablets in Subjects With Mild (Child-Pugh: Class A), Moderate (Child-Pugh: Class B) Hepatic Impairment, and Normal Hepatic Function
Brief Title: A Study of the Pharmacokinetics and Safety of CS0159 in Subjects With Hepatic Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS0159-HI-CN-I-05
Record Dates: First submitted 2025-03-05; First posted 2025-03-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Guoup 1 (Experimental): Single oral dose of CS0159 in subjects with Child-Pugh Grade A
  Interventions: Drug: CS0159
- Guoup 2 (Experimental): Single oral dose of CS0159 in subjects with Child-Pugh Grade B
  Interventions: Drug: CS0159
- Guoup 3 (Experimental): Single oral dose of CS0159 in healthy subjects with normal liver function
  Interventions: Drug: CS0159

INTERVENTIONS:
Drug: CS0159 — Single oral dose of CS0159 4mg

SUMMARY:
Phase I Study of the Pharmacokinetics and Safety of CS0159 in Subjects With Hepatic Injury

DETAILED DESCRIPTION:
To evaluate the PK characteristics of CS0159 in subjects with mild hepatic impairment (Child-Pugh Class A), moderate hepatic impairment (Child-Pugh Class B), and sex, age, and body weight-matched healthy subjects with normal hepatic function, so as to provide a scientific basis for the appropriate dose and/or dosing interval adjustment in subjects with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign a written informed consent form, and are able to complete the entire trial process according to the trial requirements.
2. Subjects aged 18 to 75 years (inclusive) at the time of signing the informed consent form; male or female.
3. At screening, the weight of male subjects is ≥50 kg, the weight of female subjects is ≥45 kg, and both are ≤100 kg; body mass index [BMI = weight (kg)/height2 (m2)] is within 18.0-32.0 kg/m2 (inclusive).
4. Subjects and their partners agree to have no plans for conception or sperm/egg donation from the signing of the informed consent until 6 months after the last dosing of the study drug and voluntarily take effective contraception measures.

For subjects with hepatic impairment, the following inclusion criteria must also be met:

1. Group 1: subjects with mild hepatic impairment (Child-Pugh Class A, score 5-6), see Appendix 1 for specific scoring.
2. Group 2: subjects with moderate hepatic impairment (Child-Pugh Class B, score 7-9), see Appendix 1 for specific scoring.
3. Subjects with hepatic impairment caused by prior primary liver disorders, who have not used albumin within 14 days prior to screening, and have been diagnosed with stable (≥1 month) hepatic impairment through past medical history, physical examination, laboratory tests, or imaging examinations.
4. Subjects who have not taken any medications within 4 weeks prior to screening, or, for those requiring long-term treatment for hepatic impairment and/or other comorbid diseases, have been on stable medication for at least 4 weeks (stable medication is determined by the investigator, excluding medications prohibited by the protocol).

Exclusion Criteria:

1. Subjects known to have a history of allergy to components or excipients of the investigational product, those with an allergic constitution (multiple drug and food allergies), or those with a history of allergic diseases (such as asthma, urticaria, eczema dermatitis, etc.).
2. Subjects who have a malignant tumor, or a history of malignant tumor regardless of time from diagnosis.
3. Subjects with severe infection, trauma, intestinal operation, or other major surgery within 4 weeks prior to screening.
4. Subjects with a history of organic heart disease, cardiac failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, or long QT syndrome, or who have symptoms and family history of long QT syndrome (indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes).
5. Subjects who have or previously had arrhythmia that requires clinical intervention and may affect survival during the trial; or those with clinically significant electrocardiogram abnormalities at screening [such as tachycardia/bradycardia requiring drug therapy, second- to third-degree atrioventricular block, or prolonged QTcF interval (male QTcF > 450 ms, female QTcF > 470 ms) (corrected using Fridericia's formula), or other clinically significant abnormalities determined by the clinician].
6. Serum creatinine > upper limit of normal (ULN), or estimated glomerular filtration rate (eGFR) calculated using the modification of diet in renal disease (MDRD) formula ˂60 mL/min/1.73 m2.
7. Subjects who are scheduled for surgery or are likely to require hospitalization during the study period.
8. Subjects with blood pressure ≥140/90 mmHg (allow retesting 2 times).
9. Subjects with resting heart rate >100 bpm (allow retesting 2 times).
10. Subjects positive for HIV antibody (HIV-Ab) testing.
11. Within 4 weeks prior to drug dosing, subjects who have used herbal medicines or any drugs that may affect CYP3A enzyme activity (such as CYP3A inducers, i.e., barbiturates, carbamazepine, glucocorticoids, etc.; inhibitors, i.e., SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, etc.).
12. Subjects who have taken any medications (including herbal medicines, vitamins, and health supplements) within 14 days before dosing (or 5 half-lives, whichever is longer), except for stable medications in subjects with hepatic impairment.
13. Subjects who have participated in other clinical trials and received investigational products or medical devices within 1 month prior to screening, using the date of the last dosing in the clinical study as the time reference (if the clinical study drug has a long half-life, at least 5 half-lives must have elapsed between dosing in that study and dosing in this study).
14. Subjects who have experienced blood loss or blood donation of ≥400 mL within 3 months prior to dosing, or plan to donate blood within 1 month after the end of this trial.
15. Subjects who are addicted to smoking, or smoked more than 5 cigarettes per day within 3 months prior to screening, or unable to stop any tobacco product use during the study period.
16. At present or within 1 month prior to screening, subjects with regular alcohol use, that is, women who consume more than 7 units of alcohol per week, men who consume more than 14 units of alcohol per week (1 unit = 14 g of pure alcohol); or subjects who test positive for alcohol breath at baseline; or who are unable to abstain from alcohol during the study.
17. Subjects with drug abuse or use of soft drugs (e.g., marijuana) within 3 months prior to dosing, or use of hard drugs (e.g., cocaine, amphetamines, phencyclidine, etc.) within 1 year prior to dosing, or positive baseline urine drug abuse screening.
18. Subjects who have consumed foods or beverages containing grapefruit juice/pomelo juice, or containing methylxanthine purines (tea, coffee, cola, chocolate, and energy drinks) within 48 h before dosing, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.
19. Subjects who cannot tolerate venipuncture or have a fear of needles or blood.
20. Subjects who have received a vaccine injection within 1 month prior to screening.
21. Pregnant or breastfeeding women, or those with a positive blood pregnancy test.
22. Subjects who, in the investigator's opinion, have poor compliance or other factors making them unsuitable for participation in this trial.

Supplementary exclusion criteria for subjects with hepatic impairment (subjects meeting any one of the following criteria will be excluded):

1. Subjects with positive syphilis tests.
2. Subjects with a history of liver transplant.
3. Subjects with drug-induced liver injury.
4. Subjects with acute liver injury due to various causes.
5. Subjects with cholestatic liver disease.
6. Imaging indicates the presence of hepatocellular carcinoma (HCC) lesions and/or alpha-fetoprotein >20 ng/mL.
7. At screening, serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5× ULN.
8. Subjects with hepatic failure and/or advanced hepatic decompensation as evidenced by:

   1. hepatic encephalopathy grade ≥3,
   2. ascites grade ≥2, and/or
   3. portal hypertension ≥10 mmHg.
9. Apart from the primary liver disease itself, subjects with any history of serious diseases, or with a medical history or clinically significant abnormal laboratory test that the investigator believes may affect the study results, including but not limited to a history of diseases of the circulatory system, endocrine system, nervous system, digestive system, urinary system, or blood, immune, psychiatric, and metabolic diseases.

Supplementary exclusion criteria for healthy subjects with normal hepatic function (subjects meeting any one of the following criteria will be excluded):

1. Subjects positive for treponema pallidum (TP) antibody test.
2. Subjects with previous primary diseases of major organs, including but not limited to neurological/psychiatric, cardiovascular, gastrointestinal, respiratory, urinary, endocrine, hematological, immune, and other diseases, whom the investigator determines are unsuitable to participate in this trial.
3. Subjects with a history of hepatic dysfunction, or those whose results from various examinations during screening (including physical examination, vital signs, hematology, urinalysis, blood chemistry, coagulation function, thyroid function, 12-lead electrocardiogram, chest PA X-ray, abdominal ultrasound, etc.) are judged by the investigator to be abnormal and of clinical significance.
4. Subjects with an age not within ±10 years of the mean age of subjects with moderate and mild hepatic impairment, and/or weight not within ±10% of the mean weight of subjects with moderate and mild hepatic impairment.
5. Subjects with past or current hepatitis B and/or hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of CS0159 (Cmax) | Day1 to day3
  Peak concentration
Pharmacokinetic parameters of CS0159 (AUC0-t) | Day1 to day3
  Area under the concentration-time curve from time zero to the last measurable concentration
Pharmacokinetic parameters of CS0159 (AUC0-∞) | Day1 to day3
  Area under the curve from time 0 extrapolated to infinite time
Pharmacokinetic parameters of CS0159 (Tmax) | Day1 to day3
  Time to peak concentration
Pharmacokinetic parameters of CS0159 (t1/2) | Day1 to day3
  Eliminate terminal half-life
Pharmacokinetic parameters of CS0159 (CL/F) | Day1 to day3
  Apparent clearance
Pharmacokinetic parameters of CS0159 (MRT) | Day1 to day3
  Mean Residence Time
Pharmacokinetic parameters of CS0159 (Vz/F) | Day1 to day3
  (Vz/F)

SECONDARY OUTCOMES:
Safety evaluation endpoints | Baseline to Day 7
  Including the incidence and severity of AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao wei feng, Master, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality